CLINICAL TRIAL: NCT00271271
Title: Phase II Clinical Trial With the Combination Gemcitabine, Oxaliplatin and Vinorelbine as First Line Treatment in Patients With Non-small Cell Bronchopulmonary Cancer
Brief Title: Efficacy Study of GEMOX Combination and Vinorelbine in NSCL Patients
Acronym: GON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8907
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Oxaliplatin; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oxaliplatine / gemcitabine / Vinorelbine

SUMMARY:
Primary:

·To evaluate the activity of the combination of gemcitabine, oxaliplatin and vinorelbine as first line treatment in patients with non-small cell bronchopulmonary cancer

Secondary:

·To evaluate the toxicity of the combination

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell bronchopulmonary cancer established by histological and/or cytological methods;
* Advanced or metastatic disease (stage IIIB or IV);
* At least one measurable lesion with one dimension (>= 20 mm by CT scan or >=10 mm by CT scan) outside of the irradiated area;
* No prior chemotherapy;
* Previous radiotherapy permitted as long as there has been a washout period of at least 4 weeks;
* Age >= 18 years old;
* ECOG Performance Status (PS): 0-1;
* Life expectancy >3 months;
* Hepatic and renal functions and blood count satisfactory:

  * Blood counts: white blood cells >= 3.0 x 10^9/l, neutrophils >= 1.5 x 10^9/l, platelets >= 150 x 10^9/l, haemoglobin >= 9 g/dl,
  * Hepatic function: bilirubin within the limit of the normal upper value, aspartate transaminases (AST) or alanine transaminases (ALT) <= 2.5 times the normal upper value
  * Renal function: creatinine clearance (calculated according to Cockroft and Gault) >= 40 ml/min;
* Patients of reproductive age must use an effective contraceptive method;
* Informed consent form signed before any procedure undertaken connected with the study

Exclusion Criteria:

* Pregnant or breastfeeding patient;
* Past record of other cancers (excluding basocellular or epidermoid cutaneous carcinoma or cured carcinoma of the cervix);
* Symptomatic cerebral or leptomeningeal metastases;
* Symptomatic peripheral neuropathy > 1 (NCI-CTC grade);
* Presence of a serious disease or medical condition incompatible with the study (at the discretion of the investigator);
* Treatment with another test product or participation in another therapeutic trial in the 4 weeks preceding inclusion in the study;
* Concomitant treatment by any other anticancer therapy;
* Concomitant treatment with phenytoin.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-06; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Objective rate of response (ORR) according to the RECIST criterion, as evaluated by a review panel of outside experts.

SECONDARY OUTCOMES:
Progression free survival (PFS), Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France